CLINICAL TRIAL: NCT06686420
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Study, to Assess the Effect of Bifidobacterial Supplementation on Bowel Movements.
Brief Title: Investigation of the Effects of a Bifidobacterial Strain on Bowel Movement in Healthy Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Morinaga Milk Industry Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFCRO-171
Record Dates: First submitted 2024-10-28; First posted 2024-11-13 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Infrequent Bowel Movements
MeSH Terms: interventions — galacto-N-biose-lacto-N-biose I phosphorylase, Bifidobacterium longum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B. longum (Experimental): Participants will be instructed to consume the capsule containing the live B. longum strain.
  Interventions: Dietary Supplement: B. longum
- Placebo (Placebo Comparator): Participants will be instructed to consume the placebo capsule without any live bacteria.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: B. longum — On the first day of the intervention period, participants will be instructed to consume two capsules of the live B. longum strain daily with a glass of water before breakfast for the next eight weeks.
  Arms: B. longum
Dietary Supplement: Placebo — On the first day of the intervention period, participants will be instructed to consume two capsules, which are without any live bacteria, daily. They should take these before breakfast with a glass of water, for the following eight weeks.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate whether a supplement containing the B. longum strain works to alleviate constipation in adults.

The main questions it aims to answer are:

Does a supplement containing the B. longum strain increase the number of spontaneous bowel movements per week, improve stool consistency, and enhance the quality of life?

Participants will:

Take a supplement containing the B. longum strain or a placebo every day for 8 weeks.

Maintain an e-diary as per the instructions. Visit the clinic for screening assessments, baseline, and end of the intervention for stool sample submission.

DETAILED DESCRIPTION:
Constipation significantly impacts the quality of life, and one of the main causes is the disruption of the gut microbiota. Probiotics have been reported to have a beneficial effect on the intestines, and Bifidobacteria, in particular, have shown functionality in relieving constipation.This randomized, placebo-controlled, clinical trial investigates the effect of Bifidobacterial supplementation intervention on bowel movement in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Is willing to participate in the study and comply with its procedures.
* Be able to give written informed consent.
* Adults aged ≥18 years and ≤65 years.
* Experience less than 3 bowel movements per week within the past three months.
* ≥25% of bowel movements with stool firmness, less than Type-3 based on Bristol Stool Scale (BSS), within the past three months.
* Record less than 6 bowel movements in eDiary App during the two-week run-in period.
* Is willing to maintain the current diet and level of physical activity throughout the study period.

Exclusion Criteria:

* Participants who are pregnant or wish to become pregnant during the study, or who are currently breastfeeding.
* Participants currently of biological childbearing potential, but not using continuous effective method of contraception, as outlined below:

  1. Complete abstinence from intercourse two weeks prior to administration of the Study Product, throughout the clinical study, until the completion of follow-up procedures or for two weeks following discontinuation of the Study Product in cases where Participant discontinues the study prematurely. (Participants utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding two weeks when they present to the clinic for the final Visit).
  2. Has a male sexual partner who is surgically sterilized prior to the Screening Visit and is the only male sexual partner for that Participant.
  3. Sexual partner(s) is/are exclusively female.
  4. Use of acceptable method of contraception, such as a spermicide, mechanical barrier (e.g., male condom, female diaphragm), tubal ligation, or contraceptive pill. The Participant must be using this method for at least one week prior to and one week following the end of the study.
  5. Use of any intrauterine device (IUD) or contraceptive implant. The Participant must have the device inserted at least two weeks prior to the first Screening Visit, throughout the study, and two weeks following the end of the study.
* Participants reporting current, or historical alcohol or drug abuse in the past year.
* Participants who have quit smoking in the 6-months prior to screening.
* Participants with a known allergy to the Study Product's active or inactive ingredients.
* Participants with chronic disease who require long-term medication throughout the whole study period.
* Participants with a significant acute, chronic or un-controlled coexisting illness or is taking medication/supplements that would put the Participant at risk or confound the interpretation of the study results, as judged by the investigator.
* Participants who regularly take medications, that are thought to affect defecation, including regular laxative use. (Occasional laxative use (PRN) < 3 times per month is acceptable).
* Participants who regularly consume supplements that are thought to affect defecation, including but not limited to fiber, iron, and magnesium.
* Participants who are consuming oral antibiotics at screening, during run-in and for the duration of the study.
* Participants who have consumed probiotic supplements and prebiotic supplements 8 weeks prior to Visit 2.
* Participants who have consumed fermented foods, that aid in bowel movement improvement such as yogurt, kefir, sauerkraut, kimchi, soy-based fermented food, miso, natto and fermented cheese, etc. within the 4 weeks prior to Visit 2.
* Participants who are diagnosed with or undergoing treatment for any gastrointestinal conditions such as coeliac disease, diarrhea, Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, gastroesophageal reflux disease (GERD) or have undergone significant gastrointestinal surgery (appendectomy allowed).
* Participants diagnosed with clinical depression, Parkinson's disease, anxiety, or an anxiety related disorder, who are undergoing treatment with medication.
* Participants with clinically significant abnormal laboratory results at screening.
* Individuals who are cognitively impaired and/or who are unable to give informed consent.
* Participants may not be participating in other clinical studies. If the participant has previously taken part in an experimental study, the Investigator must ensure sufficient time has elapsed before entry to this study to ensure the integrity of the results.
* Any Participant who is an employee of the investigational site or an Atlantia Clinical Trials employee or their close family member or a member of their household.
* Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in SBM frequency | From baseline to Week 8
  Change in mean weekly frequency of SBM, as measured by the daily bowel diary from baseline to the end of intervention. Frequency will be defined as the mean weekly number of SBM during the 2-week run-in period prior to Visit 2, for baseline, and during the final 2-week period of the intervention prior to Visit 3, for end of intervention.

SECONDARY OUTCOMES:
Change in SBM frequency | From baseline to Week 2, Week 4 and Week 6
  Change in mean weekly frequency of SBM, as measured by the daily bowel diary from baseline to Week 6. Frequency will be defined as the mean weekly number of SBM from baseline to Week 1-2, baseline to Week 3-4, baseline to Week 5-6.
Change in stool consistency | From baseline to Week 8
  Change in mean daily stool consistency as measured from the Bristol Stool Scale (BSS) in the daily bowel dairy from baseline to the end of intervention. Stool Consistency will be defined as the mean daily stool consistency during the 2-week run-in period prior to Visit 2, for baseline, and during the final 2-week period of the intervention, for end of intervention.
Patient Assessment of Constipation Symptoms (PAC-SYM) Questionnaire | From baseline to Week 4 and Week 8
  Change in self-reported constipation related symptoms as assessed by the Total Score of the Patient Assessment of Constipation Symptoms (PAC-SYM) Questionnaire.
Patient Assessment of Constipation Quality of Life (PAC-QoL) Questionnaire | From baseline to Week 4 and Week 8
  Change in self-reported impact of constipation on Quality of Life as assessed by the Total Score of the Patient Assessment of Constipation Quality of Life (PAC-QoL) Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Boetto, Principal Investigator — STTI
Locations (1):
- Atlantia Clinical Trials, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT06686420/Prot_002.pdf